CLINICAL TRIAL: NCT04136249
Title: Improvement of Neuromuscular Function, Fatigue and Quality of Life by Optimizing Muscle Building and Nutrition in Colorectal Cancer: a Pilot Study
Acronym: ColCanter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: Dr Laurent GERGELE (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-A00504-53
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2019-10

CONDITIONS: Cancer; Cachexia; Cancer
Keywords: cancer; cachexia; nutrition; physical exercice
MeSH Terms: conditions — Neoplasms; Cachexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control chimiotherapeutic arm (No Intervention): Standard care as comparaison procedure that includes chemotherapy
- Physical over-activity (Experimental): The procedure under study which includes a re-training mixing EMS and EXC with a nutrition adapted to the needs related to the physical over-activity following the chemotherapy
  Interventions: Dietary Supplement: Over physical activity

INTERVENTIONS:
Dietary Supplement: Over physical activity — 105/5000 resistance training combined with nutritional monitoring on maximum strength of knee extensors
  Arms: Physical over-activity

SUMMARY:
This study is based on the assumption that muscle strength and muscle mass will be better preserved in an "intervention" group with specific management combining retraining and nutritional monitoring compared to the "no intervention" group and that this will be positive consequences for fatigue and quality of life. In addition, this project is also based on the assumption that these gains will be at least partially preserved 3 months after the end of specific care.

DETAILED DESCRIPTION:
Cancer patients have a significant risk of losing muscle mass, mainly related to cachexia, as a result of metabolic changes associated with the tumor process and treatments. However, it is reinforced by the sedentary lifestyle that results from fatigue felt by patients. This loss of muscle mass causes in patients with general weakness and a loss of maximum strength. However, it has recently been shown that muscle weakness is not only a consequence of muscle atrophy, but also the result of contractile dysfunction, which reduces fatigue resistance to exercise. Cancer cachexia can also be directly associated with high levels of subjective cancer-related fatigue.

While it has been reported that resistance exercise programs can mitigate the deleterious effects of the disease and / or treatment, the results are likely to be partly debated because these programs are not optimized.

This study proposes to use eccentric contraction and electromyostimulation because there is evidence that the effects of these methods used in combination may be greater in developing strength and muscle mass.

In addition to muscle building, nutritional monitoring is a key element of recovery. For example, it has been shown that a preoperative exercise and nutritional support program has the potential to reduce sarcopenia and improve postoperative outcomes in elderly sarcopenic patients with gastric cancer.

Ultimately, this study is based on the assumption that muscle strength and muscle mass will be better preserved in an "intervention" group with specific management combining retraining and nutritional monitoring compared to the "no intervention" group and that this will be positive consequences for fatigue and quality of life. In addition, this project is also based on the assumption that these gains will be at least partially preserved 3 months after the end of specific care.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over 18 years old
* Patient operated on for a first colorectal cancer (adenocarcinoma) and requiring adjuvant chemotherapy
* Patient with the consent of a physician to participate in the innovative muscle building program
* Patient able to go at least once a week for 12 weeks to the Private Hospital of the Loire in Saint-Etienne (the other 2 weekly sessions that can take place in the patient's home)
* Patient affiliated or beneficiary of a social security scheme
* Patient having signed the free and informed consent

Exclusion Criteria:

* Comorbidities potentially affecting participation or test results (unstable, neuromuscular, musculoskeletal or vascular diseases affecting the lower limbs, such as radiculopathy, myopathy or neuropathy)
* Technical necessity to convert laparoscopy into laparostomy
* Patient unable to follow verbal instructions that could affect test and / or exercise procedures
* Patient participating in another clinical study
* Protected patient: major under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Pregnant, lactating or parturient woman
* Patient hospitalized without consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11-02 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Isometric force | 3 months
  This objective will be evaluated using an isometric ergometer and the force will be expressed in Newtons. This parameter will be analyzed using a mixed linear model adjusted to the group and clinically relevant factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé de la Loire 39, Saint-Étienne-de-Montluc, Pays de la Loire Region, France

IPD SHARING:
Plan to Share IPD: Undecided